CLINICAL TRIAL: NCT04332809
Title: A Randomized Controlled Trial on Irrigation of Open Appendectomy Wound With Gentamicin- Saline Solution Versus Saline Solution for Prevention of Surgical Site Infection.
Brief Title: A Randomized Controlled Trial on Wound Irrigation in Open Appendectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Associate professor of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mansoura333
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saline-gentamicin irrigation (Active Comparator): layer-by-layer irrigation of the appendectomy wound will be performed using Saline-gentamicin solution
  Interventions: Procedure: saline-gentamicin irrigation
- Saline irrigation (Active Comparator): layer-by-layer irrigation of the appendectomy wound will be performed using Saline solution
  Interventions: Procedure: saline irrigation
- No irrigation (No Intervention): ayer-by-layer irrigation of the appendectomy wound will not be performed

INTERVENTIONS:
Procedure: saline-gentamicin irrigation — Layer-by-layer irrigation of the appendectomy wound will be performed using saline-gentamicin solution
  Arms: Saline-gentamicin irrigation
Procedure: saline irrigation — Layer-by-layer irrigation of the appendectomy wound will be performed using saline solution
  Arms: Saline irrigation

SUMMARY:
A large retrospective study compared wound irrigation with antiseptic solution, with antimicrobial agent, and with normal saline in patients undergoing open appendectomy and concluded an evident superiority of antibiotic wound irrigation over both normal saline and antiseptic solution.

The present trial aimed to assess the efficacy of layer-by-layer wound irrigation with gentamicin-saline solution versus saline solution in prevention of incisional SSI after open appendectomy for acute appendicitis. We postulated that irrigation of every layer of the surgical wound separately would help reduce the incidence of incisional SSI by eradication of bacterial contamination of each layer which may occur during delivery, manipulation, and removal of the inflamed appendix through the McBurney's incision.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients of both genders aging between 16 and 65 years who presented to the emergency department with acute appendicitis. Acute appendicitis was diagnosed by clinical examination and intraoperative findings and the diagnosis was confirmed with histopathologic examination of the removed appendix.

Exclusion Criteria:

* Patients with appendicular mass, appendicular abscess, appendicitis associated with generalized peritonitis, acute abdomen due to other causes as revealed intraoperatively, patients with normal appendix as revealed intraoperatively and after histopathologic examination, patients taking long course of steroid therapy or immunosuppressive treatment, and patients unwilling to participate in the trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infection | 6 weeks after surgery
  SSI was defined according to the standard criteria devised by the center for disease and control (CDC). Purulent drainage from the wound, cellulitis requiring antibiotics, or the opening of a closed wound were considered criteria of Incisional SSI

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No